CLINICAL TRIAL: NCT04433208
Title: Dietary Study of a Complex Oligosaccharide With and Without a Probiotic in Healthy Volunteers
Brief Title: Dietary Supplement With and Without a Probiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-CT-001
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Probiotics; Histamine H2 Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Probiotic) (Experimental): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily
  Interventions: Dietary Supplement: Probiotic
- Cohort 2 (Complex oligosaccharide) (Experimental): Day 1-14: Subjects receive 18 g dose of complex oligosaccharide orally twice daily
  Interventions: Dietary Supplement: Complex oligosaccharide
- Cohort 3 (4.5 g Dose of Complex oligosaccharide + Probiotic) (Experimental): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 4.5 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 4.5 g dose of complex oligosaccharide orally twice daily
  Interventions: Dietary Supplement: Complex oligosaccharide; Dietary Supplement: Probiotic
- Cohort 4 (9 g dose of Complex oligosaccharide + Probiotic) (Experimental): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 9 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 9 g dose of complex oligosaccharide orally twice daily
  Interventions: Dietary Supplement: Complex oligosaccharide; Dietary Supplement: Probiotic
- Cohort 5 (18 g dose of Complex oligosaccharide + PPI + Probiotic +/- H2 Blocker) (Experimental): First Course Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) and PPI orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Second Course Day 29-35: Subjects receive standard probiotic dose (mixed in aqueous diluent) and may receive H2 blocker* orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 36-42: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  *4 subjects received H2 blocker, 4 subjects did not receive H2 blocker during second course
  Interventions: Dietary Supplement: Complex oligosaccharide; Dietary Supplement: Probiotic; Other: PPI; Other: H2 Blocker
- Cohort 6 (18 g dose of Complex oligosaccharide + Probiotic) (Experimental): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Interventions: Dietary Supplement: Complex oligosaccharide; Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Complex oligosaccharide — Complex oligosaccharide concentrate
  Arms: Cohort 2 (Complex oligosaccharide); Cohort 3 (4.5 g Dose of Complex oligosaccharide + Probiotic); Cohort 4 (9 g dose of Complex oligosaccharide + Probiotic); Cohort 5 (18 g dose of Complex oligosaccharide + PPI + Probiotic +/- H2 Blocker); Cohort 6 (18 g dose of Complex oligosaccharide + Probiotic)
Dietary Supplement: Probiotic — Probiotic
  Arms: Cohort 1 (Probiotic); Cohort 3 (4.5 g Dose of Complex oligosaccharide + Probiotic); Cohort 4 (9 g dose of Complex oligosaccharide + Probiotic); Cohort 5 (18 g dose of Complex oligosaccharide + PPI + Probiotic +/- H2 Blocker); Cohort 6 (18 g dose of Complex oligosaccharide + Probiotic)
Other: PPI — Over-the-counter proton pump inhibitor (PPI)
  Arms: Cohort 5 (18 g dose of Complex oligosaccharide + PPI + Probiotic +/- H2 Blocker)
Other: H2 Blocker — Over-the-counter H2 blocker
  Arms: Cohort 5 (18 g dose of Complex oligosaccharide + PPI + Probiotic +/- H2 Blocker)

SUMMARY:
Complex oligosaccharides can alter the gut microbiome by aiding in the growth of certain organisms, and possibly, inhibiting others. The synergy with a probiotic may enhance gastrointestinal colonization.

DETAILED DESCRIPTION:
The study will evaluate the synergy of the use of a complex oligosaccharide with and without a probiotic on the human microbiome in healthy volunteers. The combination should support general gastrointestinal health.

The study a multi-dose randomized cohort trial using 10 subjects per cohort for a total of 60 healthy adult volunteers ages 18-44.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-44 years
* Willingness to complete all study procedures and clinic visits, and provide required samples
* Provides informed consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding, or intend to become pregnant during the course of this study
* Subjects with history of lactose intolerance
* Subjects who are on a PPI regimen
* Subjects who have taken a probiotic during the previous 30 days, or intends to take a probiotic during the study.
* Subjects who have taken antibiotics within 120 days
* Alcohol or drug abuse during the last 12 months, including passing a screen for drugs of abuse at screening
* Unstable medical condition, in the opinion of the investigator
* Clinically significant abnormal laboratory test results at screening
* Participation in a clinical research trial within 30 days prior to screening
* Unable to give informed consent
* Any condition which may preclude subject's ability to comply with and complete the study or may pose a risk to the health of the subject

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 4.5 g dose of complex oligosaccharide orally twice daily Day 8-14:Subjects receive only 4.5 g dose of complex oligosaccharide orally twice daily
Period: Overall Study
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Started | 10 | 10 | 10 | 10 | 12 | 10
Completed | 10 | 9 | 9 | 10 | 10 | 8
Not Completed | 0 | 1 | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic): Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 9 g dose of complex oligosaccharide orally twice daily Day 8-14:Subjects receive only 9 g dose of complex oligosaccharide orally twice daily
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 12 | 10 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 12 | 10 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7) | 34.6 (4.4) | 31.7 (8.2) | 34.1 (6.4) | 31.1 (6.9) | 34.6 (5.8) | 33.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 4 | 4 | 2 | 26
  Male | 5 | 5 | 4 | 6 | 8 | 8 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 3 | 3 | 4 | 2 | 19
  Not Hispanic or Latino | 10 | 3 | 7 | 7 | 8 | 8 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 2 | 2 | 1 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 1 | 3 | 3 | 2 | 15
  White | 0 | 5 | 6 | 4 | 6 | 5 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 2 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 12 | 10 | 62
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14.2 (2.45) | 14.3 (1.88) | 13.7 (1.51) | 14.2 (1.62) | 14.8 (1.40) | 14.6 (1.31) | 14.3 (1.69)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Levels of B.Infantis in Stool by Quantitative PCR
Description: qPCR analysis uses primers for species and strain on DNA extracted from stool samples and is reported as genome copies per nanogram of DNA. The higher the value, the greater indication of engraftment of B.infantis signal over time indicating retention of introduced species.
Time Frame: All Cohorts - Day 1, 5, 8, 15 and 29; Cohort 5 - additionally Days 33, 36, 43, 50 and 57
Population: Changes in microbiome species abundance and diversity
Measure: Geometric Mean (95% Confidence Interval); unit: copies/ng DNA
Groups:
- Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker): First Course Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) and PPI orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Second Course Day 29-35: Subjects receive standard probiotic dose (mixed in aqueous diluent) and may receive H2 blocker* orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 36-42: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  *4 subjects received H2 blocker, 4 subjects did not receive H2 blocker during second course
  Complex oligosaccharide: Complex oligosaccharide concentrate
  Probiotic: Probiotic
  PPI: Over-the-counter proton pump inhibitor (PPI)
  H2 Blocker: Over-the-counter H2 blocker
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10 | 9
copies/ng DNA
  Day 1 | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33]
  Day 5: number analyzed (Participants) | 10 | 8 | 10 | 9 | 10 | 9
  Day 5 | 322.38 [180.53 to 575.66] | 3.33 [3.33 to 3.33] | 127.48 [25.63 to 634.11] | 64.03 [11.95 to 343.12] | 263.20 [63.06 to 1098.58] | 371.37 [38.92 to 3543.55]
  Day 8 | 276.67 [120.16 to 637.05] | 3.33 [3.33 to 3.33] | 271.21 [70.59 to 1042.03] | 180.24 [65.35 to 497.154] | 391.72 [23.31 to 6581.70] | 1454.29 [103.68 to 20398.61]
  Day 15 | 5.36 [1.83 to 15.67] | 3.33 [3.33 to 3.33] | 21.83 [2.78 to 171.51] | 18.89 [1.87 to 190.47] | 111.46 [4.98 to 2494.13] | 1636.68 [64.35 to 41626.43]
  Day 22: number analyzed (Participants) | 10 | 9 | 9 | 10 | 10 | 8
  Day 22 | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 9.13 [2.16 to 38.63]
  Day 29: number analyzed (Participants) | 10 | 9 | 9 | 10 | 10 | 8
  Day 29 | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33] | 3.33 [3.33 to 3.33]
  Day 33: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 33 |  |  |  |  | 59.74 [9.24 to 386.15] |
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 36 |  |  |  |  | 72.34 [8.26 to 633.77] |
  Day 43: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 43 |  |  |  |  | 22.96 [1.25 to 421.63] |
  Day 50: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 50 |  |  |  |  | 4.07 [2.59 to 6.41] |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0
  Day 57 |  |  |  |  | 3.33 [3.33 to 3.33] |
Statistical Analysis 1: Comparison: Cohort 1 (Probiotic) vs Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) vs Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic); Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Changes in Concentration of Blood Parameters From Day 1 to Day 15
Description: Blood samples are collected and tested for analysis of the levels of cytokines using Luminex-based chemistry to assess for immunology screening and safety monitoring of liver function, renal function, and electrolytes and glucose.
Time Frame: Day 1 - 15
Population: Descriptive statistics will not include analytes that were not detected in samples or not detected at high enough concentrations to be above the lower limit of quantification. Values for analytes below the lower limit of quantification were imputed with that value for inclusion in the descriptive statistics. Measurements were only taken for Cohorts 1, 2 and 6.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Number analyzed (Participants) | 10 | 10 | 9
pg/mL
  Brain-Derived Neurotrophic Factor (BDNF) - Study Day 1 | 14.10 (5.38) | 17.36 (5.92) | 16.30 (4.51)
  Brain-Derived Neurotrophic Factor (BDNF) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Brain-Derived Neurotrophic Factor (BDNF) - Study Day 15 | 13.43 (6.06) | 16.82 (4.34) | 16.00 (3.94)
  Eotaxin-2 - Study Day 1 | 928.70 (261.85) | 1129.50 (247.49) | 1004.89 (362.32)
  Eotaxin-2 - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Eotaxin-2 - Study Day 15 | 931.80 (289.66) | 1214.00 (304.64) | 1112.78 (437.58)
  Interleukin-1 beta (IL-1 beta) - Study Day 1 | 10.90 (2.32) | 9.90 (4.22) | 9.28 (4.12)
  Interleukin-1 beta (IL-1 beta) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Interleukin-1 beta (IL-1 beta) - Study Day 15 | 9.75 (3.91) | 10.50 (4.46) | 10.68 (2.07)
  Interleukin-1 receptor antagonist (IL-1ra) - Study Day 1 | 108.80 (30.44) | 118.90 (27.52) | 108.33 (26.83)
  Interleukin-1 receptor antagonist (IL-1ra) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Interleukin-1 receptor antagonist (IL-1ra) - Study Day 15 | 118.90 (17.76) | 111.22 (36.89) | 104.00 (25.09)
  Interleukin-12 Subunit p40 (IL-12p40) - Study Day 1 | 0.66 (0.17) | 0.60 (0.17) | 0.65 (0.08)
  Interleukin-12 Subunit p40 (IL-12p40) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Interleukin-12 Subunit p40 (IL-12p40) - Study Day 15 | 0.69 (0.14) | 0.60 (0.22) | 0.67 (0.17)
  Interleukin-18 (IL-18) - Study Day 1 | 207.10 (124.68) | 208.00 (77.16) | 187.33 (79.43)
  Interleukin-18 (IL-18) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Interleukin-18 (IL-18) - Study Day 15 | 187.20 (100.18) | 223.22 (92.55) | 180.00 (85.23)
  Latency-Associated Peptide of Transforming Growth Factor beta 1 (LAP TGF-b1) - Study Day 1 | 35.20 (6.00) | 33.90 (4.91) | 30.67 (10.46)
  Latency-Associated Peptide of Transforming Growth Factor beta 1 (LAP TGF-b1) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Latency-Associated Peptide of Transforming Growth Factor beta 1 (LAP TGF-b1) - Study Day 15 | 34.70 (7.41) | 35.33 (5.89) | 32.11 (8.54)
  Macrophage Inflammatory Protein-1 beta (MIP-1 beta) - Study Day 1 | 427.80 (184.10) | 390.30 (275.65) | 329.22 (161.56)
  Macrophage Inflammatory Protein-1 beta (MIP-1 beta) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Macrophage Inflammatory Protein-1 beta (MIP-1 beta) - Study Day 15 | 430.60 (222.27) | 408.11 (295.14) | 335.44 (148.03)
  Vascular Endothelial Growth Factor (VEGF) - Study Day 1 | 288.70 (112.99) | 233.60 (79.24) | 200.11 (95.08)
  Vascular Endothelial Growth Factor (VEGF) - Study Day 15: number analyzed (Participants) | 10 | 9 | 9
  Vascular Endothelial Growth Factor (VEGF) - Study Day 15 | 303.70 (125.31) | 252.78 (117.20) | 198.22 (89.24)

3. Secondary Outcome: Summary of the Evaluation of the Use of Proton Pump Inhibitors for Protection of B. Infantis Levels in Cohorts 5 and 6 by Visit
Description: Evaluation of B. infantis levels in Dose Group 5 will be compared to B. infantis levels in Dose Groups 6 using descriptive statistics including geometric means and 95% confidence intervals of the genome copy number per nanogram of DNA (B. infantis copies/ng DNA).
Time Frame: Day 1, 5, 8, 15, 22, 29, 33, 43, 50, 57
Population: Microbiome Population (Two cohorts received 18g of HMO with B. infantis and will be distinguished from each other by one receiving the proton pump inhibitor omeprazole. In addition, the cohort dosed with omeprazole received a second round of dosing with half of the subjects receiving famotidine in addition to B. infantis and 18g of HMO and the remainder not receiving any acid reducing drugs)
Measure: Geometric Mean (95% Confidence Interval); unit: B. infantis (copies/ng DNA)
Arm/Group | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Number analyzed (Participants) | 10 | 9
B. infantis (copies/ng DNA)
  Day 1 | 3.3 [3.3 to 3.3] | 3.3 [3.3 to 3.3]
  Day 5 | 263.2 [63.1 to 1098.6] | 371.4 [38.9 to 3543.5]
  Day 8 | 391.7 [23.3 to 6581.7] | 1454.3 [103.7 to 20398.6]
  Day 15 | 111.5 [5.0 to 2494.1] | 1636.7 [64.4 to 41626.4]
  Day 22 | 3.3 [3.3 to 3.3] | 9.1 [2.2 to 38.6]
  Day 29 | 3.3 [3.3 to 3.3] | 3.3 [3.3 to 3.3]
  Day 33: number analyzed (Participants) | 10 | 0
  Day 33 | 59.7 [9.2 to 386.2] |
  Day 36: number analyzed (Participants) | 10 | 0
  Day 36 | 72.3 [8.3 to 633.8] |
  Day 43: number analyzed (Participants) | 10 | 0
  Day 43 | 23.0 [1.3 to 421.6] |
  Day 50: number analyzed (Participants) | 10 | 0
  Day 50 | 4.1 [2.6 to 6.4] |
  Day 57: number analyzed (Participants) | 10 | 0
  Day 57 | 3.3 [3.3 to 3.3] |

4. Secondary Outcome: Concentrations (µmol/g) of Lactic Acid in Stool Samples From Day 1 to Day 29
Description: Descriptive statistics including means and standard deviation of lactate (Cohort 1; 0g HMO + B. infantis, Cohort 2; 18 g HMO, engrafted subjects and not engrafted subjects from Cohorts 5 & 6 combined; 18g HMO + B.
  infantis). Descriptive statistics will not include analytes that were not detected in greater than 50% of samples.
Time Frame: Day 1, 8, 15, 29
Population: Cohort 1 (no HMO, only B. infantis), Cohort 2 (18g HMO, no B. infantis). Cohorts 5 and 6 were combined because both of these groups received 18g HMO +B. infantis and this was pre-specified in the analysis plan for this outcome. The measurement of lactic acid was expected, therefore, to be very similar between these two groups and the goal of this analysis was to compare the combination of a probiotic with complex oligosaccharides to each of these separately (Cohorts 1 and 2, respectively).
Measure: Mean (Standard Deviation); unit: µmol/g
Groups:
- Cohort 5 + Cohort 6 (Engrafted): Cohort 5:
  First Course Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) and PPI orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Second Course Day 29-35: Subjects receive standard probiotic dose (mixed in aqueous diluent) and may receive H2 blocker* orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 36-42: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  *4 subjects received H2 blocker, 4 subjects did not receive H2 blocker during second course
  Complex oligosaccharide: Complex oligosaccharide concentrate
  Cohort 6:
  Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Probiotic: Probiotic
  PPI: Over-the-counter proton pump inhibitor (PPI)
  H2 Blocker: Over-the-counter H2 blocker
  Engrafted: Subjects will be deemed "engrafted" if the B. infantis signal, as measured by qPCR, is above the limit of detection (L.O.D.) of the assay on days 5, 8, and 15
- Cohort 5 + Cohort 6 (Not Engrafted): Cohort 5:
  First Course Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) and PPI orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Second Course Day 29-35: Subjects receive standard probiotic dose (mixed in aqueous diluent) and may receive H2 blocker* orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 36-42: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  *4 subjects received H2 blocker, 4 subjects did not receive H2 blocker during second course
  Complex oligosaccharide: Complex oligosaccharide concentrate
  Cohort 6:
  Day 1-7: Subjects receive standard probiotic dose (mixed in aqueous diluent) orally once daily in combination with 18 g dose of complex oligosaccharide orally twice daily Day 8-14: Subjects receive only 18 g dose of complex oligosaccharide orally twice daily
  Not Engrafted: Subjects with no signal on any one of those days will be deemed "not engrafted" because the introduced species was not consistently retained.
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 5 + Cohort 6 (Engrafted) | Cohort 5 + Cohort 6 (Not Engrafted)
Number analyzed (Participants) | 10 | 9 | 11 | 8
µmol/g
  Lactic acid - Day 1 | 0.11 (0.04) | 0.39 (0.74) | 3.18 (10.02) | 0.14 (0.05)
  Lactic acid - Day 8 | 0.18 (0.14) | 0.20 (0.20) | 0.17 (0.05) | 0.16 (0.08)
  Lactic acid - Day 15 | 0.13 (0.11) | 0.14 (0.06) | 0.85 (1.14) | 0.12 (0.06)
  Lactic acid - Day 29 | 0.18 (0.14) | 0.13 (0.05) | 0.40 (0.93) | 0.12 (0.06)

5. Secondary Outcome: Changes in Concentration of Blood Parameters From Day 1 to Day 15 (Factor VII)
Description: as for outcome 2
Time Frame: Day 1 - 15
Population: Descriptive statistics will not include analytes that were not detected in samples or not detected at high enough concentrations to be above the lower limit of quantitation. Values for analytes below the lower limit of quantification were imputed with that value for inclusion in the descriptive statistics. Data were only available for Cohorts 1, 2 and 6.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Number analyzed (Participants) | 10 | 10 | 9
ug/mL
  Factor VII - Day 1 | 354.0 (104.0) | 382.9 (90.0) | 362.3 (76.0)
  Factor VII - Day 15 | 358.5 (124.7) | 403.6 (99.6) | 384.2 (79.5)

6. Secondary Outcome: Changes in Concentration of Blood Parameters From Day 1 to Day 15 (ICAM-1)
Description: Blood samples are collected and tested for analysis of the levels of cytokines using Luminex-based chemistry to assess for immunology screening and safety monitoring of liver function, renal function and electrolytes and glucose.
Time Frame: Day 1 - 15
Population: Descriptive statistics will not include analytes that were not detected in samples or not detected at high enough concentrations to be above the lower limit of quantification. Values for analytes below the lower limit of quantification were imputed with that value for inclusion in the descriptive statistics. Data were only available for Cohorts 1, 2 and 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
Number analyzed (Participants) | 10 | 10 | 9
ng/mL
  Intercellular Adhesion Molecule 1 (ICAM-1) - Day 1 | 71.0 (18.4) | 68.6 (23.5) | 65.1 (21.8)
  Intercellular Adhesion Molecule 1 (ICAM-1) - Day 15 | 65.2 (16.2) | 75.1 (28.6) | 73.0 (27.5)

ADVERSE EVENTS:
Time Frame: Cohort 1,2,3,4,6 - 38 days Cohort 5 - 73 days
Arm/Group | Cohort 1 (Probiotic) | Cohort 2 (Complex Oligosaccharide) | Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic) | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 2/10 | 1/10 | 2/12 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Probiotic) (N=10) | Cohort 2 (Complex Oligosaccharide) (N=10) | Cohort 3 (4.5 g Dose of Complex Oligosaccharide + Probiotic) (N=10) | Cohort 4 (9 g Dose of Complex Oligosaccharide + Probiotic) (N=10) | Cohort 5 (18 g Dose of Complex Oligosaccharide + PPI + Probiotic +/- H2 Blocker) (N=12) | Cohort 6 (18 g Dose of Complex Oligosaccharide + Probiotic) (N=10)
Bacteria Vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cubital Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT04433208/Prot_SAP_000.pdf